CLINICAL TRIAL: NCT00003171
Title: Phase II Clinical Evaluation of Bryostatin 1 in Patients With Myelodysplastic Syndrome
Brief Title: Bryostatin 1 in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065975; P30CA022453 (NIH); WSU-D-1468; NCI-T97-0047
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — bryostatin 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of bryostatin 1 in treating patients with myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of bryostatin 1 in patients with myelodysplastic syndrome. II. Determine the qualitative and quantitative toxic effects of bryostatin 1. III. Determine the duration of response and survival of patients receiving this therapy.

OUTLINE: This is a two stage study. Patients receive bryostatin 1 by continuous infusion over 72 hours every 14 days for 4 cycles. Responding patients may continue treatment in the absence of disease progression or unacceptable toxicity. Patients with complete response receive 2 additional cycles. Patients with no response receive 4 additional cycles. Patients are re-evaluated after every 4 cycles.

PROJECTED ACCRUAL: 14 to 27 patients will be accrued within 2 years into this 2 stage study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed refractory anemia, refractory anemia with excess blasts, refractory anemia with excess blasts in transformation, refractory anemia with ringed sideroblasts, or chronic myelomonocytic leukemia with significant cytopenias of at least 4 weeks duration No more than 1 prior treatment for disease Not eligible for allogeneic bone marrow transplantation if less than 60 years of age

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: Hematocrit less than 26% (or requiring transfusion) for at least 4 weeks Absolute neutrophil count less than 1000/mm3 for at least 4 weeks Platelet count less than 50/mm3 for at least 4 weeks Hepatic: Bilirubin less than 1.5 mg/dL Transaminase less than 2.5 times upper limit of normal Renal: Creatinine less than 1.5 mg/dL Creatinine clearance of at least 60 mL/min Other: Not pregnant or lactating Fertile patients must use effective contraception while on study and for 100 days afterwards No uncontrolled or life-threatening infection

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy No concurrent treatment with growth factors Chemotherapy: At least 4 weeks since prior chemotherapy (8 weeks for mitomycin or nitrosourea) and recovered Endocrine therapy: No concurrent use of steroids Radiotherapy: At least 4 weeks since prior radiation therapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05; Primary Completion 1999-07 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayad M. Al-Katib, MD, FACP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States